CLINICAL TRIAL: NCT06506435
Title: RADIOACTIVE - Radiotherapy Patient Education With Virtual Reality
Brief Title: Radiotherapy Patient Education With Virtual Reality
Acronym: RADIOACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Benjamin Rich, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240355
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Cancer
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Informational Video (Active Comparator): Participants in this group will watch a two-dimensional (2D) informational video that explains the radiation treatment process. Total participation is up to 8 weeks.
  Interventions: Behavioral: Two Dimensional (2D) Informational Video
- Virtual Reality: 1st Person Perspective (Experimental): Participants in this group will have a virtual reality experience presented from a first-person perspective. Participants will wear a Meta Quest Pro virtual reality headset, immersing themselves in a scenario that replicates the radiation treatment process. Total participation is up to 8 weeks.
  Interventions: Behavioral: First-Person Virtual Reality Video
- Virtual Reality: 3rd Person Perspective (Experimental): Participants in this group will wear a Meta Quest Pro virtual reality headset and use virtual reality to observe the radiation treatment scenario from a standing position within the room, enabling them to witness both the CT scan and radiation machine from an external viewpoint. Total participation is up to 8 weeks.
  Interventions: Behavioral: Third-Person Virtual Reality Video

INTERVENTIONS:
Behavioral: Two Dimensional (2D) Informational Video — A 30-minute informational video. The two dimensional (2D) video provides information about the radiotherapy process. Participants will receive this one-time intervention in-person, prior to treatment.
  Arms: Informational Video
Behavioral: First-Person Virtual Reality Video — A 30-minute virtual reality video, experienced through a headset, provides an immersive portrayal of the radiotherapy process from a first-person perspective. Participants will receive this one-time intervention in-person, prior to treatment.
  Arms: Virtual Reality: 1st Person Perspective
Behavioral: Third-Person Virtual Reality Video — A 30-minute virtual reality video, experienced through a headset, provides an immersive portrayal of the radiotherapy process from a third-person perspective. Participants will receive this one-time intervention in-person, prior to treatment.
  Arms: Virtual Reality: 3rd Person Perspective

SUMMARY:
The purpose of this research study is to investigate the impact of virtual reality experiences on individuals undergoing radiotherapy, aiming to assess whether this immersive technology can reduce anxiety and enhance patient overall treatment satisfaction. By comparing different virtual reality techniques and a standard informational video, the study seeks to identify optimal strategies for leveraging virtual reality to improve the patient experience during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven cancer
2. ≥18 years of age
3. Able to speak and read English and/or Spanish
4. Receiving radiotherapy at the University of Miami

Exclusion Criteria:

1. Prior radiation therapy
2. Pregnant or nursing women
3. Men or women of childbearing potential who are unwilling to employ adequate contraception
4. Patients unable to consent or are prisoners
5. Participants with impaired decision-making capacity
6. Any serious illness or medical condition that would compromise patient safety during virtual reality as judged by the treating physician
7. Unwilling or unable to watch virtual reality video
8. Unwilling to fill out survey forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Level of Anxiety measured by scores on the State-Trait Anxiety Inventory (STAI) | Baseline, up to 2 weeks
  The State-Trait Anxiety Inventory (STAI) is a brief and widely used self-assessment tool validated to measure anxiety in individuals undergoing medical therapy or other stressful experiences. The scale consists of 20 items, with separate scales for trait and state. Scores on the Likert scale, ranging from 0 to 4, provide an assessment of symptom severity in patients dealing with various medical conditions (state) as well as baseline status (trait). Higher scores indicate higher levels of anxiety.

SECONDARY OUTCOMES:
Change in Level of Anxiety measured by scores on the State-Trait Anxiety Inventory (STAI) | Baseline, up to 8 weeks
  The State-Trait Anxiety Inventory (STAI) is a brief and widely used self-assessment tool validated to measure anxiety in individuals undergoing medical therapy or other stressful experiences. The scale consists of 20 items, with separate scales for trait and state. Scores on the Likert scale, ranging from 0 to 4, provide an assessment of symptom severity in patients dealing with various medical conditions (state) as well as baseline status (trait). Higher scores indicate higher levels of anxiety.
Change in Radiation Oncology Knowledge Assessment Survey (ROKAS) | baseline, up to 1 day (after intervention)
  Radiation Oncology Knowledge Assessment Survey (ROKAS) is a questionnaire designed to evaluate patient understanding of the radiotherapy treatment process. It consists of questions tailored to assess knowledge related to radiation therapy, including about procedures and potential side effects associated with treatment. ROKAS score ranges from 0-11 with higher scores indicating higher knowledge of radiation oncology.
Change in Health-Related Quality of Life measured by the Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire | Baseline, up to 8 weeks
  The absolute difference score on the FACT-G will be compared between the arms. The FACT-G is a 27-item questionnaire that covers four health-related quality of life (HR-QOL) sub-domains: physical, social, emotional, and functional well-being. Each of the questions will be scored on a scale from 0 (Not at all) to 4 (Very much) using a manual scoring template in which some items are reverse scored. Higher scored indicate better HR-QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Rich, MD, Principal Investigator — University of Miami; Crystal Chen, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No